CLINICAL TRIAL: NCT06564259
Title: The Relationship Between Serum Beta-2 Microglobulin (sB2M) Levels and CD8+ Cell Infiltration in Hodgkin Lymphoma Tissues: Impact on Chemotherapy Outcomes
Brief Title: Relationship Between Serum β2-Microglobulin and Infiltration of CD8+ in the Tumor Tissue of Hodgkin's Lymphoma Patients
Status: Completed | Type: Observational
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Other Study IDs: 1839
Record Dates: First submitted 2024-08-18; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hodgkin Lymphoma
Keywords: serum Beta-2 Microglobulin, CD8+ cells, Hodgkin lymphoma, Predictive value, Chemotherapy.
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor lymph nodes embedded in paraffin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In newly diagnosed Hodgkin lymphoma patients, pre-treatment Beta-2 Microglobulin (B2M) levels will be measured. A thorough baseline assessment will be performed using CT imaging, and tumor tissue samples will be collected for Immunohistochemical (IHC) analysis to quantify CD8+ cell infiltration. Patients will be closely monitored throughout their treatment, with a follow-up CT scan at the end of therapy to evaluate therapeutic response. This study aims to investigate the correlation between pre-treatment B2M levels and CD8+ immune cell infiltration in tumor tissues, assessing their potential as predictive markers for chemotherapy response.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with Hodgkin lymphoma
* No prior history of malignancy
* Absence of primary or secondary immunodeficiencies

Exclusion Criteria:

* Patients who have previously undergone treatment
* Patients with acute or chronic infections
* Patients with renal disorders
* Individuals with autoimmune diseases
* HIV-positive patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included a cohort of 144 patients newly diagnosed with Hodgkin lymphoma. Patients were between the ages of 14 and 71 years, with an almost balanced representation of both genders. All participants had a confirmed Hodgkin lymphoma diagnosis based on histopathological examination. The study population reflected a diverse range of disease stages and subtypes, providing a comprehensive understanding of the relationship between pre-treatment Beta-2 Microglobulin (B2M) levels, CD8+ cell infiltration, and chemotherapy response in this patient population.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Therapeutic response | 2-4 months
  Achieving complete remission after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Firas Hussien, Prof., Study Chair — Tishreen University; Maram Bilal, Prof., Study Director — Tishreen University; Hasan Khalil, Ms, Principal Investigator — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code